CLINICAL TRIAL: NCT03036631
Title: Ideal Sedation for Stroke Thrombectomy
Acronym: ISST
Status: Completed | Type: Observational
Sponsor: Dr. M. Asif Taqi (Other)
Responsible Party: Sponsor-Investigator, Dr. M. Asif Taqi, Director Neuroendovascular, Neurovascular Research Foundation
Organization: Neurovascular Research Foundation (Other)
Other Study IDs: 20150455
Record Dates: First submitted 2016-12-28; First posted 2017-01-30 (Estimated); Last update posted 2018-07-19 (Actual); Status verified 2018-07

CONDITIONS: Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Conscious Sedation/Monitored Anesthesia Care
- General Anesthesia

SUMMARY:
The Ideal Sedation for Stroke Thrombectomy (ISST) registry will answer the key questions whether sedation with intubation and paralytics is feasible and whether it delays the time to recanalization in comparison with conscious sedation alone. As a pilot registry, it is anticipated to enroll 40 acute stroke patients requiring mechanical thrombectomy over 12-18 months. Following enrollment, data will be collected prospectively from medical records and from patients' visits.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Suitable for intra-arterial treatment for acute stroke up to 8 hours from onset of symptoms
* Clinical equipoise for best mode of sedation

Exclusion Criteria:

* Any known allergy to either proposed medication and its alternative
* Any patient that has been intubated prior to randomization
* Posterior circulation strokes
* Age ≤ 18
* Pregnant female

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients underwent mechanical thrombectomy at Los Robles hospital, Thousand Oaks, CA
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2016-10; Primary Completion 2018-03 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
Time interval between groin puncture and final recanalization | 6 months or at study completion

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad A Taqi, Principal Investigator — Neurovascular Research Foundation
Locations (1):
- Los Robles Hospital and Medical Center, Thousand Oaks, California, United States

REFERENCES:
- [Derived] Taqi MA, Suriya SS, Sodhi A, Quadri SA, Farooqui M, Zafar A, Mortazavi MM. Ideal sedation for stroke thrombectomy: a prospective pilot single-center observational study. Neurosurg Focus. 2019 Feb 1;46(2):E16. doi: 10.3171/2018.11.FOCUS18522. PMID 30717046